CLINICAL TRIAL: NCT04492566
Title: Supervised Safety and Feasibility Evaluation of the Zone-MPC Control Algorithm Integrated Into the iAPS in Pregnant Patients With Type 1 Diabetes With Extension Into Outpatient at Home
Brief Title: Automated Insulin Delivery in Pregnant Patients With Type 1 Diabetes With Extension Into Outpatient at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sansum Diabetes Research Institute (Other)
Collaborators: Mayo Clinic (Other); Harvard University (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G200099/S001
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Results first posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Type 1 Diabetes; Pregnancy
Keywords: type 1 diabetes; pregnancy; artificial pancreas; automated insulin delivery
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- AID Evaluation (Experimental): After completing a 1-2 week CGM run-in period, subjects will complete a 48-60 hour closed-loop (CL) session in a supervised outpatient environment with medical staff present.
  For subjects who wish to continue use of the system, they will be offered the option of continuing use of the system at home in an extension phase, for the rest of their pregnancy.
  Interventions: Device: Automated Insulin Delivery

INTERVENTIONS:
Device: Automated Insulin Delivery — Participants will use the Automated Insulin Delivery (AID) iAPS system for 48-60 hours in a medically supervised session.
  For subjects who wish to continue use of the system, they will be offered the option of continuing use of the system at home in an extension phase, for the rest of their pregnancy.
  Other Names: Interoperable Artificial Pancreas System (iAPS)

SUMMARY:
This clinical trial is a safety and feasibility study to assess the performance of an artificial pancreas (AP) system using the Zone Model Predictive control (Zone-MPC) and Health Monitoring System (HMS) algorithms embedded into the iAPS platform for pregnant patients with type 1 diabetes (T1D).

DETAILED DESCRIPTION:
The system will be evaluated on up to 21 pregnant adult subjects with type 1 diabetes age 18-45 years old at three clinical sites (Sansum Diabetes Research Institute, Mayo Clinic Rochester MN and Mt Sinai Hospital, New York City). Subjects will complete a 48-60 hour closed-loop (CL) session in a supervised outpatient environment with medical staff present. During the session, subjects will bolus for all meals and snacks, and will perform their usual daily activities while being accompanied by study medical staff.

For subjects who wish to continue use of the system, they will be offered the option of continuing use of the system at home in an extension phase, for the rest of their pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 45 years at the time of screening.
* Clinical diagnosis of type 1 diabetes
* Currently using an insulin pump at the time of screening.
* HbA1c ≤ 9%, as performed by point of care or central laboratory testing.
* Pregnant 14+0/7 to 32+6/7 weeks gestation.
* Singleton pregnancy without any other significant known complications, such as preeclampsia, premature rupture of membranes, 2nd/3rd trimester bleeding, fetal growth or fluid abnormalities.
* No proven or suspected fetal malformations diagnosed in the current pregnancy.
* Bolus for all meals and snacks that contain ≥ 5 grams of carbohydrate.
* Willing to switch to, or continue Novolog or Humalog for the closed-loop session.
* Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial.
* Willing to abide by the study protocol and use study-provided devices.
* Have a care partner with the following responsibilities: knowing subject whereabouts and being promptly available for contact by study staff during the day and night, residing in the same dwelling as subject during the night, being agreeable to all device training during the supervised HCL session and additional training on hyper- and hypoglycemia treatment, and assisting with emergency care if needed, such as transportation to the hospital or emergency department.

Exclusion Criteria:

* Known unstable cardiac disease or untreated cardiac disease, as revealed by history or physical examination.
* Concurrent use of Afrezza or any non-insulin glucose-lowering agent other than metformin (including GLP-1 agonists, Pramlintide, DPP-4 inhibitors, SGLT-2 inhibitors, sulfonylureas).
* Hemophilia or any other bleeding disorder
* Prior history of Preterm Premature Rupture of Membranes (PPROM)
* Significant hyperemesis interfering with carbohydrate intake
* Laboratory results:

  1. A1C > 9%
  2. Abnormal liver or renal function (Transaminase >2 times the upper limit of normal, creatinine > 1.5 mg/dL)
  3. Liver and renal function testing drawn at screening visit or within three months prior to screening (for other purposes) will suffice for enrollment purposes
* Dermatological conditions that would preclude wearing a CGM sensor or infusion site.
* Any condition that could interfere with participating in the trial, based on investigator judgment.
* Participation in another pharmaceutical or device trial at the time of enrollment or during the study.
* Having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial
* History of severe hypoglycemia in the past 6 months
* History of DKA requiring hospitalization in the past 6 months
* Significant chronic kidney disease (eGFR < 60) or hemodialysis
* Significant liver disease
* History of adrenal insufficiency
* History of abnormal TSH consistent with hypothyroidism or hyperthyroidism that is not appropriately treated
* History of high dose steroid use in the past 8 weeks

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Dassau, PhD, Principal Investigator — Harvard University John A Paulson School of Engineering and Applied Sciences; Yogish Kudva, MD, Principal Investigator — Mayo Clinic; Carol Levy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Barak Rosenn, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Grenye O'Malley, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Kristin Castorino, DO, Principal Investigator — Sansum Diabetes Research Institute; Jordan Pinsker, MD, Principal Investigator — Sansum Diabetes Research Institute
Locations (3):
- United States (3):
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - Mayo Clinic, Rochester, Minnesota
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Levy CJ, Kudva YC, Ozaslan B, Castorino K, O'Malley G, Kaur RJ, Levister CM, Church MM, Desjardins D, McCrady-Spitzer S, Ogyaadu S, Trinidad MC, Reid C, Rizvi S, Deshpande S, Zaniletti I, Kremers WK, Pinsker JE, Doyle FJ, Dassau E; LOIS-P Diabetes and Pregnancy Consortium. At-Home Use of a Pregnancy-Specific Zone-MPC Closed-Loop System for Pregnancies Complicated by Type 1 Diabetes: A Single-Arm, Observational Multicenter Study. Diabetes Care. 2023 Jul 1;46(7):1425-1431. doi: 10.2337/dc23-0173. PMID 37196353
- [Result] Ozaslan B, Levy CJ, Kudva YC, Pinsker JE, O'Malley G, Kaur RJ, Castorino K, Levister C, Trinidad MC, Desjardins D, Church MM, Plesser M, McCrady-Spitzer S, Ogyaadu S, Nelson K, Reid C, Deshpande S, Kremers WK, Doyle FJ , III, Rosenn B, Dassau E. Feasibility of Closed-Loop Insulin Delivery with a Pregnancy-Specific Zone Model Predictive Control Algorithm. Diabetes Technol Ther. 2022 Jul;24(7):471-480. doi: 10.1089/dia.2021.0521. Epub 2022 Apr 26. PMID 35230138

RESULTS

PARTICIPANT FLOW:
Groups:
- AID Evaluation: After completing a 1-2 week CGM run-in period, subjects will complete a 48-60 hour closed-loop (CL) session in a supervised outpatient environment with medical staff present.
  For subjects who wish to continue use of the system, they will be offered the option of continuing use of the system at home in an extension phase, for the rest of their pregnancy.
  Automated Insulin Delivery: Participants will use the Automated Insulin Delivery (AID) iAPS system for 48-60 hours in a medically supervised session.
  For subjects who wish to continue use of the system, they will be offered the option of continuing use of the system at home in an extension phase, for the rest of their pregnancy.
Period: Overall Study
Arm/Group | AID Evaluation
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Ten participants were enrolled in the study and used the system from their enrollment until delivery of the baby.
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Glycated Hemoglobin [Mean (Standard Deviation); unit: percentage of glycated hemoglobin] | 5.8 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Time in Target Glucose Range
Description: Time in target glucose range 63-140 mg/dL measured by CGM to determine safety and efficacy of the integrated system
Time Frame: Duration of iAPS Use During Pregnancy up to 40 weeks of Use
Measure: Mean (Standard Deviation); unit: percent time
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
percent time | 78.6 (9.2)

2. Secondary Outcome: Overnight Time in Target Glucose Range
Description: Sensor glucose time within the target range of 63-140 mg/dl overnight
Time Frame: Duration of iAPS Use During Pregnancy up to 40 weeks of Use
Measure: Mean (Standard Deviation); unit: percent time
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
percent time | 84.8 (7.7)

3. Secondary Outcome: Postprandial Time in Target Glucose Range
Description: Sensor glucose time within the target range of 63-140 mg/dl postprandially within 2 hours following meals and 2 hours following meals
Time Frame: Duration of iAPS Use During Pregnancy up to 40 weeks of Use
Measure: Mean (Standard Deviation); unit: percent time
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
percent time | 73.4 (11)

4. Secondary Outcome: Glucose < 63 mg/dL
Description: Percent time CGM glucose < 63 mg/dL
Time Frame: Duration of iAPS Use During Pregnancy up to 40 weeks of Use
Measure: Median (Inter-Quartile Range); unit: percent time
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
percent time | 1.6 [1.4 to 2.1]

5. Secondary Outcome: Glucose < 54 mg/dL
Description: Percent time CGM glucose < 54 mg/dL
Time Frame: Duration of iAPS Use During Pregnancy up to 40 weeks of Use
Measure: Median (Inter-Quartile Range); unit: percent time
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
percent time | 0.4 [0.3 to 0.4]

6. Secondary Outcome: Glucose > 140 mg/dL
Description: Percent time GGM glucose > 140 mg/dL
Time Frame: Duration of iAPS Use During Pregnancy up to 40 weeks of Use
Measure: Mean (Standard Deviation); unit: percent time
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
percent time | 19.7 (9.5)

7. Secondary Outcome: Glucose > 180 mg/dL
Description: Percent time GGM glucose > 180 mg/dL
Time Frame: Duration of iAPS Use During Pregnancy up to 40 weeks of Use
Measure: Median (Inter-Quartile Range); unit: percent time
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
percent time | 3.4 [3.0 to 8.0]

8. Secondary Outcome: Hypoglycemic Events Per Week
Description: Number of hypoglycemic events per week, defined as time <54 mg/dL for 15 consecutive minutes followed by time >70 mg/dL for 15 consecutive minutes.
Time Frame: Duration of iAPS Use During Pregnancy up to 40 weeks of Use
Measure: Mean (Standard Deviation); unit: events per week
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
events per week | 0.7 (0.6)

9. Secondary Outcome: Severe Hypoglycemic Events
Description: Number of hypoglycemic events that events that require active assistance of another individual
Time Frame: Duration of iAPS Use During Pregnancy up to 40 weeks of Use
Measure: Mean (Standard Deviation); unit: Number of Events
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
Number of Events | 0 (0)

10. Secondary Outcome: Hyperglycemic Events
Description: Number of episodes with ketones >1 mmol/L
Time Frame: Duration of iAPS Use During Pregnancy up to 40 weeks of Use
Measure: Mean (Standard Deviation); unit: Number of Events
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
Number of Events | 0.2 (0.42)

11. Secondary Outcome: Glucose > 250 mg/dL
Description: Percent time GGM glucose > 250 mg/dL
Time Frame: Duration of iAPS Use During Pregnancy up to 40 weeks of Use
Measure: Median (Inter-Quartile Range); unit: percent time
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
percent time | 0.2 [0.1 to 0.6]

12. Secondary Outcome: Serious Adverse Events (SAE)
Description: The total number of serious adverse events during the clinical trial
Time Frame: Duration of iAPS Use During Pregnancy up to 40 weeks of Use
Measure: Number; unit: Events
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
Events | 0

13. Secondary Outcome: Serious Adverse Device Events (SADE)
Description: The total number of serious adverse events related to the study device use during the clinical trial
Time Frame: Duration of iAPS Use During Pregnancy up to 40 weeks of Use
Measure: Number; unit: Events
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
Events | 0

14. Secondary Outcome: Adverse Device Effects (ADE)
Description: The total number of adverse device effects (ADE) during the clinical trial
Time Frame: Duration of iAPS Use During Pregnancy up to 40 weeks of Use
Population: Infusion Set Failure
Measure: Number; unit: Events
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
Events | 2

15. Secondary Outcome: Unanticipated Adverse Device Effects (UADE)
Description: The total number of unanticipated adverse device effects (UADE) during the clinical trial
Time Frame: Duration of iAPS Use During Pregnancy up to 40 weeks of Use
Measure: Number; unit: Events
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
Events | 0

16. Secondary Outcome: Mean CGM Glucose Level
Description: Mean CGM glucose level during AID use
Time Frame: Duration of iAPS Use During Pregnancy up to 40 weeks of Use
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
mg/dL | 115.1 (10.6)

17. Other Pre Specified Outcome: Closed-Loop Active Time
Description: Percent time (hours/day) of closed-loop use during the clinical trial
Time Frame: Duration of iAPS Use During Pregnancy up to 40 weeks of Use
Measure: Mean (Standard Deviation); unit: percent time
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
percent time | 94.1 (4.2)

18. Other Pre Specified Outcome: Sensor Use Time
Description: Percent Time CGM during the clinical trial
Time Frame: Duration of iAPS Use During Pregnancy up to 40 weeks of Use
Measure: Mean (Standard Deviation); unit: percent time
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
percent time | 98.5 (0.6)

19. Other Pre Specified Outcome: Maternal Outcomes: Gestational Hypertension
Description: Number of subjects who develop gestational hypertension during pregnancy
Time Frame: Duration of iAPS Use During Pregnancy up to 40 weeks of Use
Measure: Count of Participants; unit: Participants
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
Participants | 1

20. Other Pre Specified Outcome: Maternal Outcomes: Pre-eclampsia
Description: Number of subjects who develop pre-eclampsia during pregnancy
Time Frame: Duration of iAPS Use During Pregnancy up to 40 weeks of Use
Measure: Count of Participants; unit: Participants
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
Participants | 0

21. Other Pre Specified Outcome: Maternal Outcomes: Eclampsia
Description: Number of subjects who develop eclampsia during pregnancy
Time Frame: Duration of iAPS Use During Pregnancy up to 40 weeks of Use
Measure: Count of Participants; unit: Participants
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
Participants | 0

22. Other Pre Specified Outcome: Maternal Outcomes: Oligo/Polyhydramnios
Description: Number of subjects who develop oligo/polyhydramnios during pregnancy
Time Frame: Duration of iAPS Use During Pregnancy up to 40 weeks of Use
Measure: Count of Participants; unit: Participants
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
Participants | 0

23. Other Pre Specified Outcome: Maternal Outcomes: Pre Term Labor
Description: Number of subjects who develop pre term labor during pregnancy
Time Frame: Duration of iAPS Use During Pregnancy up to 40 weeks of Use
Measure: Count of Participants; unit: Participants
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
Participants | 0

24. Other Pre Specified Outcome: Maternal Outcomes: Primary Caesarian Section
Description: Number of subjects who underwent primary caesarian section
Time Frame: Duration of iAPS Use During Pregnancy up to 40 weeks of Use
Measure: Count of Participants; unit: Participants
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
Participants | 3

25. Other Pre Specified Outcome: Fetal Outcomes: Large for Gestational Age
Description: Number of infants born large for gestational age
Time Frame: At Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
Participants | 3

26. Other Pre Specified Outcome: Fetal Outcomes: Neonatal Hypoglycemia
Description: Number of infants who develop neonatal hypoglycemia. Neonatal hypoglycemia is defined as treatment requiring IV dextrose, treatment of the newborn with glucose gel is also reported, however protocols for use of glucose gel varied by delivery location.
Time Frame: At delivery and up to 48 hours afterwards
Population: No IV glucose was given, all treated with glucose gel.
Measure: Count of Participants; unit: Participants
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
Participants | 3

27. Other Pre Specified Outcome: Fetal Outcomes: Neonatal Intensive Care Unit Admission
Description: Number of infants who are admitted to the neonatal intensive care unit
Time Frame: At delivery and up to 7 days afterwards
Measure: Count of Participants; unit: Participants
Arm/Group | AID Evaluation
Number analyzed (Participants) | 10
Participants | 1

ADVERSE EVENTS:
Time Frame: Pregnancy through delivery, up to 40 weeks.
Arm/Group | AID Evaluation
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AID Evaluation (N=10)
ketosis (Endocrine disorders) | 2 (2)
COVID-19 (Infections and infestations) | 2 (2)
gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 1 (1)
exacerbation of pre-pregnancy hypertension (Pregnancy, puerperium and perinatal conditions) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/66/NCT04492566/Prot_002.pdf
  • Informed Consent Form (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/66/NCT04492566/ICF_001.pdf